CLINICAL TRIAL: NCT03069859
Title: Prophylactic Use of Tranexamic Acid for Preventing Postpartum Hemorrhage: A Randomized, Double-blinded, Placebo-controlled Pilot Trial
Brief Title: Use of TXA to Prevent Postpartum Hemorrhage
Acronym: TAPPH-1
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 418-2016
Record Dates: First submitted 2017-02-06; First posted 2017-03-03 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Post Partum Hemorrhage
Keywords: Post partum hemorrhage; Tranexamic acid; Spontaneous vaginal delivery; C-section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TXA (1g) (Experimental): For vaginal, TXA (1g) will be administered upon delivery of the anterior shoulder. For c-section, TXA (1g) will be administered when the obstetrician begins to cleanse the incision site
  Interventions: Drug: TXA (1g)
- Placebo (0.9% saline) (Placebo Comparator): For vaginal, placebo (0.9% saline) will be administered upon delivery of the anterior shoulder. For c-section, placebo (0.9% saline) will be administered when the obstetrician begins to cleanse the incision site
  Interventions: Drug: Placebo (0.9% saline)

INTERVENTIONS:
Drug: TXA (1g) — 1 gram of TXA (10 mL) diluted into 0.9% saline, 50 ml mini-bag (a total of 60 mL)
  Other Names: TXA
  Arms: TXA (1g)
Drug: Placebo (0.9% saline) — 0.9% saline (10 mL), diluted into 0.9% saline, 50 ml mini-bag (a total of 60 mL)
  Other Names: Placebo
  Arms: Placebo (0.9% saline)

SUMMARY:
Postpartum hemorrhage (PPH) occurs in up to one in ten deliveries worldwide and is the leading cause of maternal morbidity and mortality. In developing countries 30% of women develop PPH because access to a number of treatments is not readily available. Interestingly, the rate of PPH and consequently of maternal morbidity has increased significantly even in developed nations, such as Canada, over the past decades. This rate is also increasing amongst parturients in Ontario. Unfortunately, few effective preventative treatments exist.

Antifibrinolytic drugs are routinely used to reduce bleeding and the requirement for blood transfusions in a wide range of hemorrhagic conditions. The most commonly used antifibrinolytic drug is tranexamic acid (TXA). TXA is safe, affordable, with very few side effects. The World Health Organization recommended that TXA be used to reduce blood loss in several conditions, including in patients with established PPH refractory to conventional therapy.However, little is known about the prophylactic use of TXA to prevent PPH.

DETAILED DESCRIPTION:
This pragmatic, singlecentered, doubleblinded, randomized-controlled pilot trial will assess the feasibility of administering a prophylactic dose of TXA to prevent the onset of PPH amongst parturients undergoing cesarean section and spontaneous vaginal delivery. Our primary outcome will be to determine the proportion of patients who receive the investigational product successfully. Our secondary outcomes include 1) additional feasibility endpoints; 2) safety endpoints and 3) various other clinical endpoints. These clinical endpoints include a) incidence of PPH (and severe PPH); b) total number of transfusions; c) use of uterotonic drugs; and d) hospital length of stay. The investigators anticipate that TXA can be safely administered to parturients prior to delivery. The investigators also believe it will be an effective prophylactic therapy for PPH and will reduce its severity and associated morbidity. Results from this trial will be used to design and conduct a larger multicentered trial, powered to assess the outcomes of interest. Furthermore, this prophylactic use of TXA for PPH could improve outcomes of parturients not only in Ontario but worldwide where effective management of PPH remains an ongoing challenge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Singleton pregnancy
* Confirmed pregnancy
* Gestational age >32^0/7 weeks

Exclusion Criteria:

* Lack of patient consent
* Multiple pregnancy
* History of eclampsia or preeclampsia in current pregnancy
* Imminent Delivery as suspected by any RN or MD involved in delivery care
* History of cardiovascular complications:

  * Coronary artery disease or myocardial infarction
  * Repaired or unrepaired congenital heart disease
  * Vascular disease(s)
  * Severe unstable arrhythmia (e.g. Rapid atrial fibrillation, paroxysmal fibrillation, atrial flutter, etc.)
  * Congestive heart failure
* Contraindication to TXA:

  * History of venous thromboembolism
  * Active thromboembolic disease
  * High risk of thrombosis (e.g. Factor V Leiden or Protein C deficiency)
  * Acquired disturbances of colour vision
  * Allergy to TXA
  * History of seizure disorder
  * Pre-existing hematuria
  * History of renal insufficiency
* Unlikely to comply with follow-up (e.g. no fixed address, plans to move out of town)
* Prisoner status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients receiving study intervention | At time of delivery
  Proportion of patients receiving study intervention (IP) after randomization

SECONDARY OUTCOMES:
Duration of study to recruit 58 participants | Up to 4 months
  Total time required to recruit and randomize 58 patients
Proportion of budget needed to recruit 58 participants | Up to 4 months
  Cost required to recruit and randomize 58 patients
Composite number of clinical events | At 6 week (+/- 14 days) and 12 week (+/- 14 days) follow-ups assessments
  Clinical events (adverse events) such as thrombotic complications, acute renal failure, seizure, not related to a diagnosis of preeclampsia or eclampsia, receipt of mechanical ventilation and ICU admission, death, minor side effects, thrombotic complications (as listed above) in the newborn, rates of acute renal failure in the newborn, seizures in the newborn at 24-48 hours will be documented to assess for the overall safety of this trial
Incidence of PPH in study participants | Up to 4 months
  Incidence of PPH or severe PPH in study participants

CONTACTS AND LOCATIONS:
Overall Officials: Asim Q Alam, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Stephen Choi, MD,FRCPC,MSc, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin: Clinical Management Guidelines for Obstetrician-Gynecologists Number 76, October 2006: postpartum hemorrhage. Obstet Gynecol. 2006 Oct;108(4):1039-47. doi: 10.1097/00006250-200610000-00046. PMID 17012482
- [Background] Mpemba F, Kampo S, Zhang X. Towards 2015: post-partum haemorrhage in sub-Saharan Africa still on the rise. J Clin Nurs. 2014 Mar;23(5-6):774-83. doi: 10.1111/jocn.12126. Epub 2013 Mar 8. PMID 23472972
- [Background] Alam A, Choi S. Prophylactic Use of Tranexamic Acid for Postpartum Bleeding Outcomes: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Transfus Med Rev. 2015 Oct;29(4):231-41. doi: 10.1016/j.tmrv.2015.07.002. Epub 2015 Jul 17. PMID 26282735
- [Background] Carroli G, Cuesta C, Abalos E, Gulmezoglu AM. Epidemiology of postpartum haemorrhage: a systematic review. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):999-1012. doi: 10.1016/j.bpobgyn.2008.08.004. Epub 2008 Sep 25. PMID 18819848
- [Background] Calvert C, Thomas SL, Ronsmans C, Wagner KS, Adler AJ, Filippi V. Identifying regional variation in the prevalence of postpartum haemorrhage: a systematic review and meta-analysis. PLoS One. 2012;7(7):e41114. doi: 10.1371/journal.pone.0041114. Epub 2012 Jul 23. PMID 22844432
- [Background] Ford JB, Roberts CL, Simpson JM, Vaughan J, Cameron CA. Increased postpartum hemorrhage rates in Australia. Int J Gynaecol Obstet. 2007 Sep;98(3):237-43. doi: 10.1016/j.ijgo.2007.03.011. Epub 2007 May 4. PMID 17482190
- [Background] Joseph KS, Rouleau J, Kramer MS, Young DC, Liston RM, Baskett TF; Maternal Health Study Group of the Canadian Perinatal Surveillance System. Investigation of an increase in postpartum haemorrhage in Canada. BJOG. 2007 Jun;114(6):751-9. doi: 10.1111/j.1471-0528.2007.01316.x. PMID 17516968
- [Background] Mehrabadi A, Hutcheon JA, Lee L, Liston RM, Joseph KS. Trends in postpartum hemorrhage from 2000 to 2009: a population-based study. BMC Pregnancy Childbirth. 2012 Oct 11;12:108. doi: 10.1186/1471-2393-12-108. PMID 23057683
- [Background] Mehrabadi A, Liu S, Bartholomew S, Hutcheon JA, Kramer MS, Liston RM, Joseph KS; Maternal Health Study Group of the Canadian Perinatal Surveillance System (Public Health Agency of Canada). Temporal trends in postpartum hemorrhage and severe postpartum hemorrhage in Canada from 2003 to 2010. J Obstet Gynaecol Can. 2014 Jan;36(1):21-33. doi: 10.1016/S1701-2163(15)30680-0. PMID 24444284
- [Background] Knight M, Callaghan WM, Berg C, Alexander S, Bouvier-Colle MH, Ford JB, Joseph KS, Lewis G, Liston RM, Roberts CL, Oats J, Walker J. Trends in postpartum hemorrhage in high resource countries: a review and recommendations from the International Postpartum Hemorrhage Collaborative Group. BMC Pregnancy Childbirth. 2009 Nov 27;9:55. doi: 10.1186/1471-2393-9-55. PMID 19943928
- [Background] Mehrabadi A, Hutcheon JA, Lee L, Kramer MS, Liston RM, Joseph KS. Epidemiological investigation of a temporal increase in atonic postpartum haemorrhage: a population-based retrospective cohort study. BJOG. 2013 Jun;120(7):853-62. doi: 10.1111/1471-0528.12149. Epub 2013 Mar 6. PMID 23464351
- [Background] Sentilhes L, Lasocki S, Ducloy-Bouthors AS, Deruelle P, Dreyfus M, Perrotin F, Goffinet F, Deneux-Tharaux C. Tranexamic acid for the prevention and treatment of postpartum haemorrhage. Br J Anaesth. 2015 Apr;114(4):576-87. doi: 10.1093/bja/aeu448. Epub 2015 Jan 8. PMID 25571934
- [Background] Kirigia JM, Oluwole D, Mwabu GM, Gatwiri D, Kainyu LH. Effects of maternal mortality on gross domestic product (GDP) in the WHO African region. Afr J Health Sci. 2006 Jan-Jun;13(1-2):86-95. doi: 10.4314/ajhs.v13i1.30821. PMID 17348747
- [Background] Guerriero C, Cairns J, Perel P, Shakur H, Roberts I; CRASH 2 trial collaborators. Cost-effectiveness analysis of administering tranexamic acid to bleeding trauma patients using evidence from the CRASH-2 trial. PLoS One. 2011 May 3;6(5):e18987. doi: 10.1371/journal.pone.0018987. PMID 21559279
- [Background] Hoylaerts M, Lijnen HR, Collen D. Studies on the mechanism of the antifibrinolytic action of tranexamic acid. Biochim Biophys Acta. 1981 Feb 18;673(1):75-85. No abstract available. PMID 7193484
- [Background] Ker K, Edwards P, Perel P, Shakur H, Roberts I. Effect of tranexamic acid on surgical bleeding: systematic review and cumulative meta-analysis. BMJ. 2012 May 17;344:e3054. doi: 10.1136/bmj.e3054. PMID 22611164
- [Background] Perel P, Ker K, Morales Uribe CH, Roberts I. Tranexamic acid for reducing mortality in emergency and urgent surgery. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD010245. doi: 10.1002/14651858.CD010245.pub2. PMID 23440847
- [Background] Elwatidy S, Jamjoom Z, Elgamal E, Zakaria A, Turkistani A, El-Dawlatly A. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2577-80. doi: 10.1097/BRS.0b013e318188b9c5. PMID 19011538
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Novikova N, Hofmeyr GJ. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD007872. doi: 10.1002/14651858.CD007872.pub2. PMID 20614466
- [Background] Simonazzi G, Bisulli M, Saccone G, Moro E, Marshall A, Berghella V. Tranexamic acid for preventing postpartum blood loss after cesarean delivery: a systematic review and meta-analysis of randomized controlled trials. Acta Obstet Gynecol Scand. 2016 Jan;95(1):28-37. doi: 10.1111/aogs.12798. Epub 2015 Nov 12. PMID 26698831
- [Background] Shakur H, Elbourne D, Gulmezoglu M, Alfirevic Z, Ronsmans C, Allen E, Roberts I. The WOMAN Trial (World Maternal Antifibrinolytic Trial): tranexamic acid for the treatment of postpartum haemorrhage: an international randomised, double blind placebo controlled trial. Trials. 2010 Apr 16;11:40. doi: 10.1186/1745-6215-11-40. PMID 20398351
- [Background] Sentilhes L, Daniel V, Darsonval A, Deruelle P, Vardon D, Perrotin F, Le Ray C, Senat MV, Winer N, Maillard F, Deneux-Tharaux C. Study protocol. TRAAP - TRAnexamic Acid for Preventing postpartum hemorrhage after vaginal delivery: a multicenter randomized, double-blind, placebo-controlled trial. BMC Pregnancy Childbirth. 2015 Jun 14;15:135. doi: 10.1186/s12884-015-0573-5. PMID 26071040
- [Background] Nilsson IM. Clinical pharmacology of aminocaproic and tranexamic acids. J Clin Pathol Suppl (R Coll Pathol). 1980;14:41-7. No abstract available. PMID 7000846
- [Background] Deneux-Tharaux C, Sentilhes L, Maillard F, Closset E, Vardon D, Lepercq J, Goffinet F. Effect of routine controlled cord traction as part of the active management of the third stage of labour on postpartum haemorrhage: multicentre randomised controlled trial (TRACOR). BMJ. 2013 Mar 28;346:f1541. doi: 10.1136/bmj.f1541. PMID 23538918
- [Background] Tan J, Chen H, Liu Q, Chen C, Huang W. A meta-analysis of the effectiveness and safety of using tranexamic acid in primary unilateral total knee arthroplasty. J Surg Res. 2013 Oct;184(2):880-7. doi: 10.1016/j.jss.2013.03.099. Epub 2013 Apr 25. PMID 23643299
- [Background] Wesley MC, Pereira LM, Scharp LA, Emani SM, McGowan FX Jr, DiNardo JA. Pharmacokinetics of tranexamic acid in neonates, infants, and children undergoing cardiac surgery with cardiopulmonary bypass. Anesthesiology. 2015 Apr;122(4):746-58. doi: 10.1097/ALN.0000000000000570. PMID 25585004
- [Background] Grassin-Delyle S, Tremey B, Abe E, Fischler M, Alvarez JC, Devillier P, Urien S. Population pharmacokinetics of tranexamic acid in adults undergoing cardiac surgery with cardiopulmonary bypass. Br J Anaesth. 2013 Dec;111(6):916-24. doi: 10.1093/bja/aet255. Epub 2013 Jul 23. PMID 23880099
- [Background] Shimizu K, Toda Y, Iwasaki T, Takeuchi M, Morimatsu H, Egi M, Suemori T, Suzuki S, Morita K, Sano S. Effect of tranexamic acid on blood loss in pediatric cardiac surgery: a randomized trial. J Anesth. 2011 Dec;25(6):823-30. doi: 10.1007/s00540-011-1235-z. Epub 2011 Sep 24. PMID 21947753
- [Background] Faraoni D, Willems A, Melot C, De Hert S, Van der Linden P. Efficacy of tranexamic acid in paediatric cardiac surgery: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2012 Nov;42(5):781-6. doi: 10.1093/ejcts/ezs127. Epub 2012 Apr 24. PMID 22531271
- [Background] Gilad O, Merlob P, Stahl B, Klinger G. Outcome following tranexamic acid exposure during breastfeeding. Breastfeed Med. 2014 Oct;9(8):407-10. doi: 10.1089/bfm.2014.0027. Epub 2014 Jul 15. PMID 25025926
- [Derived] Alam AQ, Barrett J, Callum J, Kaustov L, Au S, Fleet A, Kiss A, Choi S. Tranexamic acid for the prevention of postpartum haemorrhage: the TAPPH-1 pilot randomized trial and lessons learned for trials in Canadian obstetrics. Sci Rep. 2023 Mar 18;13(1):4512. doi: 10.1038/s41598-023-30947-8. PMID 36934142
- [Derived] Alam A, Bopardikar A, Au S, Barrett J, Callum J, Kiss A, Choi S. Protocol for a pilot, randomised, double-blinded, placebo-controlled trial of prophylactic use of tranexamic acid for preventing postpartum haemorrhage (TAPPH-1). BMJ Open. 2017 Oct 11;7(10):e018586. doi: 10.1136/bmjopen-2017-018586. PMID 29025850